CLINICAL TRIAL: NCT05194488
Title: Evolving Treatment Modalities for Management of Patients Suffering From Disc Displacement With Reduction (A Randomized Clinical Trial)
Brief Title: Evolving Treatment Modalities for Management of Patients Suffering From Disc Displacement With Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 00010556
Record Dates: First submitted 2021-12-20; First posted 2022-01-18 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Temporomandibular Joint Disc Displacement, With Reduction
MeSH Terms: interventions — Low-Level Light Therapy; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low level laser therapy (Experimental)
  Interventions: Device: Low level laser therapy
- Botulinum toxin type A (Experimental)
  Interventions: Drug: Botulinum toxin type A
- Anterior repositioning appliance (Active Comparator)
  Interventions: Device: Anterior repositioning appliance

INTERVENTIONS:
Device: Low level laser therapy — Patients will receive low-level laser therapy on the temporomandibular joint disc
  Other Names: LLLT
  Arms: Low level laser therapy
Drug: Botulinum toxin type A — Patients will receive Botulinum toxin type A injection into the lateral pterygoid muscle under Electromyography (EMG) guidance.
  Other Names: Botox
  Arms: Botulinum toxin type A
Device: Anterior repositioning appliance — Patients will receive hard maxillary anterior repositioning appliance.
  Arms: Anterior repositioning appliance

SUMMARY:
Aim of the current study is to compare the efficacy of Low Level Laser, Botulinum toxin type A, and repositioning appliance in management of reduced temporomandibular joint disc.

ELIGIBILITY:
Inclusion Criteria:

* TMJ with audible and palpable click.
* Patients with anterior disc displacement as detected by MRI.
* Presence of full or nearly full complement of natural teeth.

Exclusion Criteria:

* Patients who have radiographic evidence of degenerative conditions of TMJ.
* Patients who have anterior disc dislocation without reduction.
* Previous history of TMD treatment.
* History of recent trauma.
* The presence of systemic diseases (i.e. rheumatoid arthritis, osteoarthritis).
* Inability or unwillingness to undergo magnetic resonance imaging (MRI) such as implanted electronic devices.
* Pregnant and lactating females.
* Patients with known allergy to botulinum toxin type A.
* Patients suffering from neurological disorders.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Temporomandibular joint dysfunction | 3 months
  Using Helkimo Anamnestic Index that includes 5 items, each having 3 possible answers scored 0, 1 or 5. The 1st item assesses limitations in range of jaw movement & is divided to 4 sections: maximum mouth opening, protrusion & lateral shift. For mouth opening , value of >40mm scores 0, 30-39mm scores 1 & <30mm scores 5. Protrusion & lateral shifts score 0 if the measurement is ≥7mm, 1 if ranging between 4-6mm and 5 if it is <4mm. These sections are added together to get a total that scores 0 if the sum of the 4 sections is 0, 1 if the subtotal is between 1-4 & 5 if the subtotal is >4. The 2nd item evaluates joint alterations that produce deviations, sounds and joint locks. The 3rd item evaluates pain when performing movements. The 4th item evaluates masticatory muscles pain. The 5th item evaluates pain on palpation in the prearticular area of TMJ. The 5 items are added and scored; 0: no TMJ involvement, 1-9: mild involvement, 10-19: moderate involvement & 20-25: severe involvement
Pain level | 3 months
  This will be assessed using the visual analogue scale (VAS) with score ranges from 0 (lowest) to 10 (highest). Higher scores indicate greater pain levels.
Temporomandibular joint clinical evaluation | 3 months
  Magnetic Resonance Imaging (MRI) will be performed for all patients using a 3 Tesla MRI scanner with a head coil. Gradient T2 (T2*) and proton-density (PD) weighted spin echo (SE) sequences will be carried out in closed and open mouth positions in the oblique sagittal plane. MRI is considered the gold standard (objective) in imaging the soft tissue components of the TMJ.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam M Bahgat, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Nermeen A Rady, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Ahmed M Abdelhamid, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Rady NA, Bahgat MM, Abdel-Hamid AM. Promising minimally invasive treatment modalities for symptomatic temporomandibular joint disc displacement with reduction: a randomized controlled clinical trial. BMC Oral Health. 2022 Dec 1;22(1):547. doi: 10.1186/s12903-022-02579-3. PMID 36456937